CLINICAL TRIAL: NCT07365657
Title: Subject-specific Finite Element Modelling of Le Fort I Osteotomy Fixation : Patient-specific Implants vs Miniplates
Brief Title: Finite Element Modelling of Le Fort I Osteotomy Fixation : PSI vs Miniplates
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 26IUFC01
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type II maloclusion: 2 patients : one with type II maloclusion, one with type III maloclusion who previously undergone orthognathic surgery
  Interventions: Other: In silico orthognathic surgery with customized implants digital only on 3D scanners
- Type III maloclusion: 2 patients : one with type II maloclusion, one with type III maloclusion who previously undergone orthognathic surgery
  Interventions: Other: In silico orthognathic surgery with customized implants digital only on 3D scanners

INTERVENTIONS:
Other: In silico orthognathic surgery with customized implants digital only on 3D scanners — 2 patients : one with type II maloclusion, one with type III maloclusion who previously undergone orthognathic surgery

SUMMARY:
This study aimed to evaluate the biomechanical performance of patient-specific versus conventional fixation for Le Fort I osteotomy using subject-specific finite element models derived from real surgical plans. Two distinct clinical scenarios-a minor advancement without impaction and a moderate advancement with posterior impaction-were analyzed to determine how surgical movements influence implant stress, bone stress, and maxillary micromotion. By combining surgical planning with validated computational modeling, this work provides clinically relevant insight to optimize PSI design and guide fixation strategy selection in orthognathic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient operated on By Pr SAVOLDELLI.
* Patient undergoing patient-specific orthognathic surgery.
* Access to numerical (digital) planning.

Exclusion Criteria:

* Previous maxillo-facial trauma.
* Facial cleft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2 patients : one with type II maloclusion, one with type III maloclusion who previously undergone orthognathic surgery
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-01-23 (Estimated); Study Completion 2026-01-23 (Estimated)

PRIMARY OUTCOMES:
Plate stress levels | At the inclusion
  assessed by FORGE software

SECONDARY OUTCOMES:
Stress on bone | At the inclusion
  Mechanical stress in mecanics is measured in Pa (Pascal)
Maxillary displacement | At the inclusion
  Displacement levels in mecanics is measured in millimeters or micrometers.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nice, Nice, Alpes Maritimes, France